CLINICAL TRIAL: NCT06443060
Title: The Effect of Virtual Reality and Buzzy Application on Pain, Fear and Anxiety During Prick Test in Children: Randomized Controlled Study
Brief Title: The Effect of Virtual Reality and Buzzy Application on Pain, Fear and Anxiety During Prick Test in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FundaTEZ
Record Dates: First submitted 2024-05-16; First posted 2024-06-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pain; Fear; Anxiety; Children, Only; Virtual Reality
Keywords: BUZZY; Virtual Reality; Pain; Fear; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Group (Experimental): After the scales are filled in, the child will be shown a cartoon film deemed appropriate by the experts by wearing VR glasses and headphones before the Prick test (average 2 minutes). The appropriate cartoon will be shown to the VR glasses group for an average of 15 minutes. After the child starts watching the cartoon, the child will be asked to extend his/her left arm and the prick test process will begin.
  Interventions: Behavioral: Virtual Reality Group
- Buzzy Application Group (Experimental): The CFS-D scale will be completed only by the child to measure the anxiety level before the procedure. To assess pain and fear, the WB-FACES pain scale and the CFS fear scale will be completed by the child, parent and researcher before the procedure. The buzzy cold and vibration device will be connected to the children in the buzzy experimental group 5-10 seconds before the procedure, at least 8-10 cm above the area to be treated (upper part of the left arm antecubital fossa) and the prick test application will be started.
  Interventions: Behavioral: Buzzy Application Group
- Control Group (Active Comparator): Children in this group will be given routine explanations according to the outpatient clinic procedure and prick test will be applied before the procedure.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Virtual Reality Group — Before starting the Prick procedure, the child in the virtual reality group, which is determined by randomisation, will be given a brief information about how the allergy test will be performed and about virtual reality. Before the Prick test (approximately 2 minutes before the Prick test), the child will start to watch a film deemed appropriate by the experts by wearing virtual reality and headphones. After the child starts watching the film, the child will be asked to extend his/her left arm and solutions will be dripped on the forearm and the puncture will be performed with a lancet. The child will continue to watch the film during the whole procedure.
  Arms: Virtual Reality Group
Behavioral: Buzzy Application Group — Before starting the prick procedure, the child in the buzzy group, which was determined by randomisation, will be given a brief information about how the allergy test will be performed and the buzzy device. The children in the buzzy experimental group will be connected to the buzzy cold and vibration device at least 8-10 cm above the area to be treated (upper part of the left arm antecubital fossa) 5-10 seconds before starting the procedure and the prick test application will be started.
  Arms: Buzzy Application Group
Other: Control Group — Before starting the prick procedure, the children in the control group determined by randomisation will be given routine explanations according to the outpatient clinic procedure before starting the procedure and the prick test will be applied.
  Arms: Control Group

SUMMARY:
Allergy is a hypersensitivity reaction to a triggering agent. Tests used in allergy are divided into two: in vivo and in vitro. Among the in vivo tests routinely used, epidermal, intradermal and patch tests are used, and the most commonly used is the skin prick test. In order to prevent the negative effects of pain, it is important to be informed about the appropriate approach to children, newborns and babies, and effective pain management, according to their cognitive development levels. Pain management in children should be done appropriately with accurate assessment tools. This will increase the quality of life, reduce hospitalizations, shorten the length of hospital stay and reduce costs. Pain experiences experienced during childhood will cause later pain experiences to be perceived as more severe and cause anxiety and fear. Anxiety is a psychological, physiological and behavioral state that develops in response to a perceived or existing threat. Anxiety, which can also be expressed as worry or anxiety, is a emotional state that can occur in various ways, such as restlessness, tension, easy fatigue, lack of concentration, muscle tension, and sleep disturbance, in which autonomic and somatic symptoms occur in the body, without any reason.

Virtual reality provides multi-sensory information as children focus on the simulated world. Virtual reality, one of the cognitive methods; It can create an environment where three-dimensional pictures or animations created on the computer can interact in people's minds. It is also defined as a distraction method created by software, which creates the feeling that users are in the environment even though they are not in the real environment, and can interact with people in the environment. When all these studies were examined, no three-group study was found comparing a distracting method with a physical method for the 7-10 age group. Additionally, there is a study that used virtual reality in the prick test, but there is no method that has been proven to be superior to virtual reality. In this study, it will be investigated whether virtual reality and buzzy applications have a reducing effect on pain, fear and anxiety compared to the control group. Virtual reality and buzzy techniques will also be compared with each other. Since no such study has been found in the literature, it is thought to contribute to the field.

DETAILED DESCRIPTION:
Allergy is a hypersensitivity reaction to a triggering agent. Tests used in allergy are divided into two: in vivo and in vitro. Among the in vivo tests routinely used, epidermal, intradermal and patch tests are used, and the most commonly used is the skin prick test. In order to prevent the negative effects of pain, it is important to be informed about the appropriate approach to children, newborns and babies, and effective pain management, according to their cognitive development levels. Pain management in children should be done appropriately with accurate assessment tools. This will increase the quality of life, reduce hospitalizations, shorten the length of hospital stay and reduce costs. Pain experiences experienced during childhood will cause later pain experiences to be perceived as more severe and cause anxiety and fear. Anxiety is a psychological, physiological and behavioral state that develops in response to a perceived or existing threat. Anxiety, which can also be expressed as worry or anxiety, is a emotional state that can occur in various ways, such as restlessness, tension, easy fatigue, lack of concentration, muscle tension, and sleep disturbance, in which autonomic and somatic symptoms occur in the body, without any reason.

Virtual reality provides multi-sensory information as children focus on the simulated world. Virtual reality, one of the cognitive methods; It can create an environment where three-dimensional pictures or animations created on the computer can interact in people's minds. It is also defined as a distraction method created by software, which creates the feeling that users are in the environment even though they are not in the real environment, and can interact with people in the environment.

When all these studies were examined, no three-group study was found comparing a distracting method with a physical method for the 7-10 age group. Additionally, there is a study that used virtual reality in the prick test, but there is no method that has been proven to be superior to virtual reality. In this study, it will be investigated whether virtual reality and buzzy applications have a reducing effect on pain, fear and anxiety compared to the control group. Virtual reality and buzzy techniques will also be compared with each other. Since no such study has been found in the literature, it is thought to contribute to the field.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between the ages of 7-10
* It will be the first time that a prick test will be applied.
* The child can speak and understand Turkish comfortably
* He and his family agree to participate in the study.
* Not having used analgesic medication at least six hours ago

Exclusion Criteria:

* The child has any diagnosed psychiatric disorder
* Having visual, auditory or speech disorders
* Having a chronic disease other than allergy

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 111 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
The Child Anxiety Scale-Stability Scale (CAS-D) | six month
  The Child Anxiety Scale-Stability Scale (CAS-D); is shaped like a thermometer with a light bulb at the bottom and horizontal lines at intervals going upwards. In this scale for children aged four to ten, children are instructed to 'Imagine that all your anxious or nervous feelings are at the bulb or bottom of the thermometer'. A transparent metre is placed over the child's rating on which ½ point increments are marked, then the ½ point increment is rounded up to the nearest number. The score can range from 0-10. Above 5 points indicates high anxiety. The CVI is 0.89, the correlation coefficient is 0.99.
Child Fear Scale (CFS) | six month
  Child Fear Scale; This scale assesses pain-related fear in children. The Child Fear Scale (CFS) developed by McMurty et al. (2011) is a scale suitable for the 5-10 age group and consists of five drawn facial expressions ranging from neutral expression (0=no fear) to frightened face (4=severe fear). It can be easily assessed by researchers and health professionals who provide care/intervention to children (McMurtry et al., 2011). There is no gold standard self-report scale that assesses fear for children. Test-retest method was used in the validity study of the scale. The Turkish version of the scale was adapted by Özalp Gerçeker et al. (2018) and the Content Validity Index (CVI) was found to be 0.89 and the correlation coefficient was 0.96 (Özalp Gerçeker et al., 2018).
Wong-Baker FACES Pain Rating Scale (WB-FACES) | six month
  Wong-Baker FACES Pain Rating Scale (WB-FACES); It was developed by Wong and Baker in 1981 and revised in 1983. It is used to diagnose pain in children and adolescents aged 3-18 years. This scale, which can be used safely over the age of three, consists of six facial parts scored between 0-10. The face shape representing no pain is evaluated as 0 points and the face shape representing severe pain is evaluated as 10 points. Participants are asked to choose the best facial expression that best describes them. WB_FACES is a scale suitable for use in Turkey (Sahiner & Bal, 2015) and will be evaluated by the parents and the researcher as well as the child's self-report in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Geçkil, Principal Investigator — Necmettin Erbakan Üniversitesi Hemşirelik Fakültesi

IPD SHARING:
Plan to Share IPD: No
After the research is over